CLINICAL TRIAL: NCT01718392
Title: Rehabilitation in Multiple Sclerosis: Influence of Exercise on Development of Insulin Resistance, Muscle Power and Aerobic Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Bert Op't Eijnde, Professor, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CME 2011/311
Record Dates: First submitted 2012-10-23; First posted 2012-10-31 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Sclerosis
Keywords: combined training; insulin resistance
MeSH Terms: conditions — Multiple Sclerosis; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Training (Experimental): 24 weeks combined exercise programme (supervised)
  Interventions: Behavioral: Training
- Control (No Intervention): sedentary/habitual lifestyle

INTERVENTIONS:
Behavioral: Training
  Other Names: 24 weeks combined exercise programma (supervised)
  Arms: Training

SUMMARY:
the purpose of this study is to investigate the development of insulin resistance in multiple sclerosis patients + explaining the effects of a combined training programme on insulin resistance, muscle power and aerobic capacity in multiple sclerosis patients

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed MS according to the McDonald criteria
* Expanded Disability Status Scale (EDSS) between 0.5 and 6
* Be able to train 5 times in 2 weeks at the University

Exclusion Criteria:

* Comorbidities like cardiovascular-, respiratory-, orthopaedic or metabolic diseases (like diabetes type 2)
* Having had an relapse in a period of 3 months prior to the start of the intervention period
* Having an relapse during the intervention period
* Pregnancy and other contra indications for physical activity
* Mental disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity (insulin profile) | change from baseline to 24 weeks
  glucose and insulin concentration measurements in blood

SECONDARY OUTCOMES:
aerobic capacity | change from baseline to 24 weeks
  by means of a submaximal endurance test (ergometer)
aerobic capacity - lactate concentrations | change from baseline to 24 weeks
  by means of a submaximal endurance test (ergometer) to determine lactate concentrations (mmol/L)
cytokine profile | change from baseline to 24 weeks
  measurements of blood cytokine levels
walking performance | change from baseline to 24 weeks
  Walking performance will be assessed by means of 2 and 6 minute walk test, 25-foot walk test, Chair rise test, Stair climb test
Self-reported measures | Change from baseline to 24 weeks
  The self-reported measures contains some questionnaires
body composition | Change from baseline to 24 weeks
  Weight, body fat% and lean tissue% will be assessed by means of a DEXA (Dual-energy X-ray absorptiometry) scan
muscle strength of knee flexor | change from baseline to 24 weeks
  by means of an isokinetic dynamometer the muscle strength and endurance will be measured
muscle strength of knee extensor | change from baseline to 24 weeks
  by means of an isokinetic dynamometer the muscle strength and endurance will be measured
muscle strength of elbow flexor | change from baseline to 24 weeks
  by means of an isokinetic dynamometer the muscle strength will be measured
muscle strength of elbow extensor | change from baseline to 24 weeks
  by means of an isokinetic dynamometer the muscle strength will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Inez Wens, M.Sc., Principal Investigator — Reval/Biomed, Hasselt University; Bert Op't Eijnde, Ph.D., Study Chair — Reval/Biomed, Hasselt University
Locations (1):
- REVAL, Diepenbeek, Belgium